CLINICAL TRIAL: NCT00293709
Title: Prospective Post Marketing Surveillance To Evaluate The Safety And Efficacy Of Etanercept Under Usual Care Settings In Patients With Psoriatic Arthritis (Psa) Treated By Dermatologists
Brief Title: Study Evaluating the Safety and Efficacy of Etanercept in Patients With Psoriatic Arthritis Treated by Dermatologists
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: 0881A6-102036; B1801126
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2014-02-26 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Arthritis, Psoriatic; Psoriasis; Skin Diseases, Papulosquamous
Keywords: Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic; Psoriasis; Skin Diseases, Papulosquamous; Arthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Psoriatic Arthritis
  Interventions: Drug: etanercept

INTERVENTIONS:
Drug: etanercept — The patients will be treated in accordance with the requirements of the labelling of Enbrel® in Germany. The dosage and duration of therapy is to be determined by the physician to meet the patients' individual needs for treatment.
  Other Names: Enbrel

SUMMARY:
The purpose of this study is to evaluate the safety profile and the effectiveness of etanercept under usual care settings in patients with PsA treated by dermatologists.

DETAILED DESCRIPTION:
Non-interventional study: subjects to be selected according to the usual clinical practice of their physician

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Psoriatic Arthritis

Exclusion Criteria:

* Sepsis or risk for sepsis,
* Acute infection,
* Hypersensitive against Etanercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients for whom the decision has already been made to initiate treatment with Enbrel® can be enrolled in this observational trial. These patients must have a proven diagnosis of Psoriatic Arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2006-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, München, Germany

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A6-102036&StudyName=Study%20Evaluating%20the%20Safety%20and%20Efficacy%20of%20Etanercept%20in%20Patients%20with%20Psoriatic%20Arthritis%20Treated%20by%20Dermatologists

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Psoriatic Arthritis: Participants with psoriatic arthritis treated by dermatologist who received etanercept (Enbrel) as per local medical practice under conditions of routine daily use, were observed for 1 year.
Period: Overall Study
Arm/Group | Participants With Psoriatic Arthritis
Started | 149
Completed | 102
Not Completed | 47
Not completed — Other | 47

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled in this study. Out of a total of 149 participants, data for baseline measure (age) was available only for 146 participants.
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 149
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 79

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and Week 52 (end of the observation period) that were absent before treatment or that worsened relative to pretreatment state. AEs included SAEs as well as non-serious AEs which occurred during the trial.
Time Frame: Baseline up to Week 52
Population: Safety analysis set included all participants who were enrolled in this study.
Measure: Number; unit: percentage of participants
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 149
percentage of participants
  AEs | 24.2
  SAEs | 1.3

2. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) Affected by Psoriasis at Week 52
Time Frame: Baseline, Week 52
Population: Efficacy analysis set included all participants who were greater than (>) 18 years of age and had confirmed diagnosis of psoriatic arthritis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Mean (Standard Deviation); unit: percentage of BSA
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 146
percentage of BSA
  Baseline (n=146) | 24.5 (22.6)
  Change at Week 52 (n=99) | -17.8 (19.6)

3. Secondary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) at Week 52
Description: PASI: combined assessment of lesion severity and area affected into single score. Body was divided into 4 sections (head, arms, trunk, and legs); each area was scored by itself and scores were combined for final PASI. For each section percent area of skin involved was estimated: 0 (0%) to 6 (90 - 100%), and severity was estimated by clinical signs: erythema, induration, and desquamation; scale: 0 (none) to 4 (maximum). Final PASI=sum of severity parameters for each section*area score*weight of section (head: 0.1, arms: 0.2, body: 0.3, legs: 0.4; total score ranged from 0 (no disease) to 72 (maximal disease).
Time Frame: Baseline, Week 52
Population: Efficacy analysis set included all participants who were >18 years of age and had confirmed diagnosis of psoriatic arthritis. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure. 'n' signifies those participants who were evaluable for this measure at given time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 143
units on a scale
  Baseline (n=143) | 15.1 (12.7)
  Change at Week 52 (n=93) | -11.8 (11.6)

4. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joints Count (DAS 28) at Week 52
Description: DAS28 calculated from the number of swollen joints (SJC) and painful joints (PJC) using the 28 joints count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 100 mm; higher scores indicated greater affectation due to disease activity). DAS28 total score range: 0-10, where DAS28 less than or equal to (=<) 3.2 = low disease activity, DAS28 >3.2 to 5.1 = moderate disease activity and >5.1 = high disease activity.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 68
units on a scale
  Baseline (n=68) | 5.1 (1.4)
  Change at Week 52 (n=43) | -2.2 (1.7)

5. Secondary Outcome: Change From Baseline in Ritchie Index at Week 52
Description: Ritchie index: the numerical measurement of joint tenderness (28 joints) in participants with arthritis. The number of quantitative evaluations of the pain experienced by the participants when the joints were subjected to firm pressure when exerted over the articular margin or in some instances by passive movement of the joint. Participant's reaction to pressure exerted by the physician were documented on 4-point scale, 0=not tender, 1=tender, 2=tender and caused wince, 3=reflexive effort to withdraw. Ritchie index was calculated as the total of the individual grades for all joints; ranged from 0 to 84, where higher score indicated higher tenderness.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 146
units on a scale
  Baseline (n=146) | 15.8 (12.8)
  Change at Week 52 (n=95) | -3.6 (20.4)

6. Secondary Outcome: Change From Baseline in Physician Global Assessment of Disease Activity at Week 52
Description: Physician global assessment of disease activity was measured on a 0 to 100 millimeter (mm) visual analog scale (VAS), with 0 mm = no disease activity to 100 mm = most possible disease activity.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 148
millimeter
  Baseline (n=148) | 60.4 (22.3)
  Change at Week 52 (n=102) | -35.8 (31.4)

7. Secondary Outcome: Number of Participants With Nail Involvement
Description: Number of participants with psoriatic arthritis affecting the nails are reported.
Time Frame: Baseline, Week 12, 52
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 147
participants
  Baseline (n=147) | 103
  Week 12 (n=131) | 81
  Week 52 (n=100) | 50

8. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Week 52
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 115
milligram per deciliter (mg/dL)
  Baseline (n=115) | 1.6 (3.0)
  Change at Week 52 (n=69) | -0.6 (3.5)

9. Secondary Outcome: Change From Baseline in Patient Assessment of Itching at Week 52
Description: Participants rated the severity of their psoriasis itching on a 0 (none) to 100 (most possible) scale.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 147
units on a scale
  Baseline (n=147) | 44.0 (29.2)
  Change at Week 52 (n=98) | -26.1 (34.2)

10. Secondary Outcome: Change From Baseline in Patient Assessment of Pain at Week 52
Description: Participants rated the severity of their psoriatic arthritis-related pain on a 0 (none) to 100 (most possible) scale.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 147
units on a scale
  Baseline (n=147) | 60.0 (27.1)
  Change at Week 52 (n=98) | -37.5 (33.8)

11. Secondary Outcome: Change From Baseline in 12-Item Short Form Health Survey (SF-12) at Week 52
Description: SF-12 questionnaire was used to determine participants' quality of life (QoL). It comprised 12 items which covered 8 concepts : physical functionality, role impairment due to physical problems, physical pain, perception of general health, vitality, social functionality, role impairment due to emotional problems, and psychological wellbeing. Results were presented in the form of 2 meta-scores, the physical component and the mental component, each ranged from 0 to 100. Higher scores=better QoL, positive changes from baseline=improvement in QoL.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Participants With Psoriatic Arthritis
Number analyzed (Participants) | 142
units on a scale
  Baseline: Physical component (n=142) | 33.5 (9.2)
  Baseline: Mental component (n=142) | 40.5 (11.5)
  Change at Week 52: Physical component (n=89) | 11.7 (10.3)
  Change at Week 52: Mental component (n=89) | 9.4 (11.9)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Participants With Psoriatic Arthritis
Serious Adverse Events (participants affected / at risk) | 2/149
Other Adverse Events (participants affected / at risk) | 34/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Psoriatic Arthritis (N=149)
Pancreatitis (Gastrointestinal disorders) | 1
Gallbladder pain (Hepatobiliary disorders) | 1
Pleural infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants With Psoriatic Arthritis (N=149)
Coronary artery disease (Cardiac disorders) | 1
Eye pain (Eye disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Stomach discomfort (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 2
Condition aggravated (General disorders) | 1
Fatigue (General disorders) | 1
Influenza like illness (General disorders) | 1
Injection site erythema (General disorders) | 2
Injection site inflammation (General disorders) | 1
Injection site pruritus (General disorders) | 2
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 2
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 2
Genital herpes (Infections and infestations) | 1
Herpes virus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 8
Oral herpes (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 1
Sinobronchitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Contusion (Injury, poisoning and procedural complications) | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase (Investigations) | 1
Arthroscopy (Investigations) | 1
Platelet count decreased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight increased (Investigations) | 1
Haemochromatosis (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 2
Alcoholism (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Ligament operation (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Transurethral prostatectomy (Surgical and medical procedures) | 1
Blood pressure fluctuation (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.